CLINICAL TRIAL: NCT04892043
Title: A Phase 1, Multicenter, Open-Label Study of SQZ-AAC-HPV as Monotherapy and in Combination With Immune Checkpoint Inhibitors in HLA-A*02+ Patients With HPV16+ Recurrent, Locally Advanced or Metastatic Solid Tumors
Brief Title: Study of SQZ-AAC-HPV in Patients With HPV16+ Recurrent, Locally Advanced or Metastatic Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Corporate Decision
Sponsor: SQZ Biotechnologies (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SQZ-AAC-HPV-101
Record Dates: First submitted 2021-04-28; First posted 2021-05-19 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Adult Solid Tumor
Keywords: solid tumors cancer; metastatic; locally advanced; cancer; cervical; head and neck; anal; penile; SQZ-AAC-HPV; HPV16; AAC; cell therapy; ipilimumab; nivolumab; checkpoint inhibitors; immunotherapy; solid tumor; HLA-A*02; therapeutic vaccine; recurrent cancer; advanced solid tumor
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms; Recurrence | interventions — Ipilimumab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1 Monotherapy Dose Escalation Phase (Experimental): In Part 1, SQZ-AAC-HPV as a monotherapy is administered every 3 weeks for up to a year.
  There are 3 groups ("Cohorts") in this Phase as follows:
  * Cohort 1a: low dose SQZ-AAC-HPV
  * Cohort 1b: high dose SQZ-AAC-HPV
  * Cohort 1c: higher or lower dose SQZ-AAC-HPV
  Interventions: Biological: SQZ-AAC-HPV
- Part 2 Combination Safety Phase (Experimental): In Part 2, SQZ-AAC-HPV in combination with immune checkpoint inhibitors (1) ipilimumab, (2) nivolumab, or (3) nivolumab plus ipilimumab is administered every 3 weeks up to a year, but the immune checkpoint inhibitors may be administered up to 2 years. There are 3 groups ("Cohorts") in this Phase as follows:
  * Cohort 2a: SQZ-AAC-HPV RP2D (Recommended Phase 2 Dose) plus ipilimumab
  * Cohort 2b: SQZ-AAC-HPV RP2D plus nivolumab
  * Cohort 2c: SQZ-AAC-HPV RP2D plus nivolumab and ipilimumab
  Interventions: Biological: SQZ-AAC-HPV; Drug: Ipilimumab; Drug: Nivolumab

INTERVENTIONS:
Biological: SQZ-AAC-HPV — Activating antigen carriers (AACs) cell therapy; therapeutic vaccine engineered from red blood cells manufactured with immunogenic epitopes of HPV16
Drug: Ipilimumab — Cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) blocking antibody
  Arms: Part 2 Combination Safety Phase
Drug: Nivolumab — Programmed cell death 1 (PD-1) blocking antibody
  Arms: Part 2 Combination Safety Phase

SUMMARY:
This is a Phase 1 open-label, multicenter study of the safety and tolerability, immunogenic effects, antitumor activity, and pharmacodynamics of SQZ-AAC-HPV as monotherapy and in combination with immune checkpoint inhibitors in HLA-A*02+ patients with recurrent, locally advanced or metastatic human papillomavirus strain 16 positive (HPV16+) solid tumors. The study includes patients with anal, rectal, cervical, head and neck, penile, vulvar, or vaginal cancer.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female patients ≥18 years of age who are HLA-A*02+ (performed during screening locally or centrally, or based on documented historic test results)
* Histologically confirmed incurable or metastatic solid tumors that are HPV16+ (performed during screening locally or centrally, or based on documented historic test results)
* Cancer must have progressed after at least 1 available standard therapy for incurable disease, or the patient is intolerant to or refuses standard therapy(ies) or has a tumor for which no standard therapy(ies) exist
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 to 1
* At least 1 measurable lesion according to RECIST 1.1
* Must have a lesion that can be biopsied with acceptable clinical risk and agree to have a fresh biopsy at Baseline and on Cycle 2 Day 8 (+/- 3 days)
* Patients must agree to venous access for the blood collection for manufacture of autologous blood product and be willing to have a central line inserted if venous access is an issue
* Adequate organ function and bone marrow reserve performed within 14 days of blood collection for manufacture of autologous blood product

Exclusion Criteria:

* Treatment with anticancer therapy, including investigational therapy, within 2 weeks prior to blood collection for manufacture of autologous blood product. For prior therapies with a half-life longer than 3 days, discontinuation of the therapy must have occurred at least 28 days prior to Cycle 1 Day 1
* Systemic treatment with either corticosteroids (>10 mg of prednisone or the equivalent per day) or other immunosuppressive medications within 14 days prior to Cycle 1 Day 1
* Patients treated with non-corticosteroid based immunosuppressive agents within the last 6 months may not be eligible and should be discussed with the Sponsor
* Patients with active, known, or suspected autoimmune disease may not be eligible and should be discussed with the Sponsor
* Patients with >Grade 1 AEs related to previous treatment with anticancer or investigational therapy that do not resolve at least 2 weeks prior to blood collection for manufacture of autologous blood product, except Grade 2 alopecia
* Known active hepatitis B or hepatitis C, or active mycobacterium tuberculosis infection
* History of any Grade 4 immune-related AE (irAE) from prior immunotherapy
* Has known active central nervous system metastases
* History of interstitial lung disease requiring steroids
* Significant acute or chronic illness
* Major surgery within 2 weeks of blood collection for manufacture of autologous blood product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-08-19 (Actual); Primary Completion 2023-11-02 (Actual); Study Completion 2023-11-02 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs; all, related, serious, and of special interest) as assessed by CTCAE version 5.0 | Up to 1 year after LPFV (Last Patient, First Visit)
  For SQZ-AAC-HPV administered as monotherapy, and in combination with immune checkpoint inhibitors (Part 1 and Part 2, respectively)
Number of participants with dose-limiting toxicity (DLT) | Through Day 28
  For SQZ-AAC-HPV as a monotherapy (Part 1)
Number of participants with DLT | Through Day 28
  For SQC-AAC-HPV in combination with immune checkpoint inhibitors (Part 2)

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Through start of a new anticancer therapy, up to 2 years after the first dose of investigational product
  Defined as the time from first dose of study treatment to first overall response of PD by RECIST v 1.1 or to death by any cause. This will be censored at the last RECIST v1.1 assessment if PD/death is not observed. For SQZ-AAC-HPV as a monotherapy, in combination with immune checkpoint inhibitors (Part 1, and Part 2, respectively).
Overall survival (OS) | Through start of a new anticancer therapy, up to 2 years after the first dose of investigational product
  Defined as the time from first dose of study treatment to death by any cause. This will be censored at the last date patient is known to be alive if death is not observed. For SQZ-AAC-HPV as a monotherapy, in combination immune checkpoint inhibitors (Part 1, and Part 2, respectively).
Objective response rate (ORR) | Through progression per RECIST v1.1 or start of new anticancer therapy, up to 2 years after first dose of investigational product
  Proportion of patients with best response of complete response [CR] and/or partial response [PR] as defined by RECIST v1.1 criteria. For SQZ-AAC-HPV as a monotherapy, in combination immune checkpoint inhibitors (Part 1, and Part 2, respectively).
Duration of Response (DoR) | Through start of a new anticancer therapy, up to 2 years after the first dose of investigational product
  Defined as the time from overall response of CR or PR to first overall response of PD by RECIST v1.1 or to death by any cause. This is defined only for patients who have a CR or PR and will be censored at the last RECIST v1.1 assessment if PD/Death is not observed. For SQZ-AAC-HPV as a monotherapy, in combination with immune checkpoint inhibitors (Part 1, and Part 2, respectively).
Best overall Response (BoR) | Through start of a new anticancer therapy, up to 2 years after the first dose of investigational product
  Evaluation of the BoR defined as CR, PR, Stable Disease [SD], Progressive Disease [PD] or Not Evaluable [NE] as defined by RECIST v1.1 criteria. For SQZ-AAC-HPV as a monotherapy, in combination with immune checkpoint inhibitors (Part 1, and Part 2, respectively).
Disease-control rate (DCR) | Through start of a new anticancer therapy, up to 2 years after the first dose of investigational product
  Proportion of patients with best response of CR or PR or SD as defined by RECIST v1.1 criteria. For SQZ-AAC-HPV as a monotherapy, in combination immune checkpoint inhibitors (Part 1, and Part 2, respectively).
Amount of investigational product (IP) from individual patient blood collection - batch yield | From leukapheresis through manufacture, a maximum of 28 days
  To determine manufacturing feasibility as assessed by batch yield (number of manufacturing runs) (Part 1)
Amount of investigational product (IP) from individual patient blood collection - product failures | From leukapheresis through manufacture, a maximum of 28 days
  To determine manufacturing feasibility as assessed by number of product failures (Part 1)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - City of Hope Medical Center, Duarte, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Oregon Health & Science University, Portland, Oregon